CLINICAL TRIAL: NCT02164760
Title: A Phase 1, Randomized, Multicentre Multinational Study to Evaluate the Safety and Feasibility of an Acellular Dermal Template Novomaix for the Treatment of Full Thickness Skin Defects in Human Patients.
Brief Title: The Safety of a Novel Acellular Dermal Template as Treatment for Burns and Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Ernst Reichmann Tissue Biology Research Unit, Zürich (Other); Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESG-09-2012; NL42113.094.12 (Other: ABR)
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Full Thickness Skin Defects
Keywords: burns; dermal substitute; scar quality; reconstruction; wound healing; wound closure
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermal substitute with STSG (Experimental): Novomaix dermal substitute in combination with STSG
  Interventions: Device: Novomaix dermal substitute in combination with STSG
- STSG alone (No Intervention): STSG alone

INTERVENTIONS:
Device: Novomaix dermal substitute in combination with STSG — Novomaix dermal substitute in combination with STSG
  Other Names: Novomaix
  Arms: Dermal substitute with STSG

SUMMARY:
In this study the safety and feasibility of an acellular dermal template (Novomaix), combined with split thickness skin grafts, for use in patients with full thickness skin defects, is tested. Results will be compared intra-patient with those obtained after conventional treatment with split thickness skin grafts. We expect this treatment to be safe, and to provide better outcome regarding scar quality.

DETAILED DESCRIPTION:
Using dermal substitutes in combination with a split-thickness skin graft (STSG) is a well acknowledged therapy in burns and reconstructive surgery. Nevertheless, the ideal substitute is not available yet. We therefore want to investigate the use of an acellular dermal template (Novomaix), in combination with STSG, to treat these defects. Adult patients with acute (burn) wounds (group 1) and scars (group 2) will be included in this study. This phase I study aims to investigate the safety and feasibility of the use of this dermal matrix, with regard to graft take, epithelialisation and complications after transplantation. Moreover, scar quality will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  1. with acute burns/trauma wounds that require skin grafting (group 1) OR
  2. with scar problems requiring surgical treatment (group 2)
* Full thickness skin defects of 50 cm2 or more, but <50% TBSA
* Skin defects must be configured in such a way that two areas of 25 cm2 can be grafted
* Informed consent by the patient

Exclusion Criteria:

* Patients with infected wounds
* Pregnant or breast feeding females
* Patients with known concomitant medical conditions that may interfere with normal wound healing (e.g. immune deficiency, HIV, diabetes, collagenoses, cancer)
* Known allergy against porcine collagen or elastin
* Patients who are expected (according to the responsible medical doctor) to be noncompliant to the study protocol. (This includes patients with severe cognitive dysfunction/impairment and severe psychiatric disorders)
* Previous enrolment of the patient into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Graft take (experimental vs control area) | 5-7 days postoperative
  Subjective assessment of two experienced observers

SECONDARY OUTCOMES:
Epithelialization | 5-7 and 18 ± 2 days days postoperative
  Subjective assessment of two experienced observers
Complication rate | Up to 12 months postoperative
  Measurement of re-operations, infection rate by culture swabs
Scar quality | 3 months
  As measured scar elasticity, scar colour and pigmentation, and a subjective scar assessment scale
Scar quality | 6 months
  As measured scar elasticity, scar colour and pigmentation, and a subjective scar assessment scale
Scar quality | 9 months
  As measured scar elasticity, scar colour and pigmentation, and a subjective scar assessment scale
Scar quality | 12 months
  As measured scar elasticity, scar colour and pigmentation, and a subjective scar assessment scale

CONTACTS AND LOCATIONS:
Overall Officials: Esther Middelkoop, Prof. dr., Principal Investigator — Red Cross Hospital
Locations (2):
- Zentrum für Schwerbrandverletzte mit Plastischer Chirurgie, Berlin, Germany
- Red Cross Hospital, Beverwijk, North Holland, Netherlands

REFERENCES:
- [Background] Boekema BK, Vlig M, Olde Damink L, Middelkoop E, Eummelen L, Buhren AV, Ulrich MM. Effect of pore size and cross-linking of a novel collagen-elastin dermal substitute on wound healing. J Mater Sci Mater Med. 2014 Feb;25(2):423-33. doi: 10.1007/s10856-013-5075-2. Epub 2013 Nov 1. PMID 24178984